CLINICAL TRIAL: NCT04783792
Title: The Effect of Phenolic Cmpounds in Osteoarthritis; a Nutritional Intervention
Brief Title: The Effect of Phenolic Compounds in Osteoarthritis; a Nutritional Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assistant Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OA supplement_( )
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Symptomatic Knee Osteoarthritis
Keywords: symptomatic knee osteoartritis, phenolic compound,
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: A randomized double-blind clinical intervention with two parallel groups lasting 3 months is proposed to elucidate the beneficial effect of a novel food supplement on OA.
  Participants will undergo clinical and biochemical testing and will provide a complete medical history and history of the disease. Demographics, smoking, alcohol consumption, eating habits and physical activity, pain, and functional inability to enroll in the study will also be recorded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ascorbic acid / phytochemical supplement (Experimental): A mixture of active phenolic compounds with ascorbic acid
  Interventions: Dietary Supplement: Ascorbic acid / phytochemical supplement
- ascorbic acid (Experimental): Ascorbic acid group
  Interventions: Dietary Supplement: Ascorbic acid

INTERVENTIONS:
Dietary Supplement: Ascorbic acid / phytochemical supplement — Ascorbic acid / phytochemical supplement
  Arms: ascorbic acid / phytochemical supplement
Dietary Supplement: Ascorbic acid — Ascorbic acid
  Arms: ascorbic acid

SUMMARY:
The main objective of the study is to elucidate the beneficial effect of a dietary supplement with phenolic compounds in patients with OA versus ascorbic acid.

The analysis of the data is expected to clarify the role of the new supplement as one with a positive effect on OA-related biomarkers, on functional abilities and on the quality of life of patients with OA.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee OA (patients with at least moderate symptoms)
* patients should be able to walk without a medical or other support device (such as a walking stick, crutches, or a kneecap).

Exclusion Criteria:

* Patients undergoing physical therapy or TENS, have rheumatoid arthritis, fibromyalgia, spinal disorders or any other disorders that according to the physician is a bias, stiffness> 30 minutes, have scheduled knee surgery or any other programmed surgery during the trial, show WOMAC pain scale <4 for pain overall, those with a diagnosis of kidney or liver disease, coagulation disorders, any form of cancer, HIV infection, type I diabetes, those with unregulated type II diabetes, those using illicit substances or having a history of substance or alcohol abuse over the past 2 years (or those who consume more than 2 typical alcoholic beverages / day in the present), those using corticosteroids within 2 months prior to randomization and during the trial, those who change their diet or supplementation 1 month or during the recruitment/trial, those using ascorbic acid supplement or any phytochemical-rich supplement, women on estrogen replacement therapy, during pregnancy or lactation and those judged by the researcher as unable to perceive and comply with the obligations laid down in the Protocol and for which consent and voluntary participation is sought.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
WOMAC™ Osteoarthritis Index Pain Subscale | 3 months
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Visual Analogue Scale - VAS | 3 months
  The Visual Analogue Scale - VAS is a unidimensional measure of pain intensity. It is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.

SECONDARY OUTCOMES:
WOMAC™ Osteoarthritis Index Stiffness Score | 3 months
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
WOMAC™ Osteoarthritis Index Physical Function Score | 3 months
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
Questionnaire SF-36 | 3 months
  SF-36 is a self-reporting set of generic, coherent, and easily administered quality-of-life measures.
Circulating Inflammatory markers | 3 months
  IL-1beta, IL-6, IL-13, TNF-alpha, endothelin
Circulating oxidative damage markers | 3 months
  MPO, oxLDL, serum oxidisability
Circulating miRNAs | 3 months
  miR-146a-5p, miR-21-5p, miR-126-3p, miR-155-5p

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Harokopio University, Athens, Attica
  - Evgenidio Hospital, Athens

IPD SHARING:
Plan to Share IPD: No